CLINICAL TRIAL: NCT03383224
Title: Angina and Genotype-Guided Smoking Cessation In PRISM-GENOMICS
Brief Title: PRISM-GENOMICS-Smoking Cessation for Patients With Coronary Artery Disease Undergoing Cardiac Catheterization or Having a Heart Attack at Barnes Hospital in St. Louis Mo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Sharon Cresci, Associate Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201412097
Record Dates: First submitted 2017-12-12; First posted 2017-12-26 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease; Smoking Cessation
Keywords: smoking cessation treatment
MeSH Terms: conditions — Coronary Artery Disease; Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Randomized to genotype-guided therapy or standard of care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Genotype-guided (A allele carriers) (Experimental): CHRNA5 rs16969968 genotype will be determined. Genotype-guided therapy will be given (A allele carriers will be given pharmacologic therapy (nicotine replacement therapy --NRT; nicotine patch used according to FDA labelling).)
  Interventions: Other: genotype-guided therapy; Drug: Nicotine patch
- Genotype-guided (GG homozygotes) (Experimental): CHRNA5 rs16969968 genotype will be determined. Genotype-guided therapy will be given (GG homozygotes will be given smoking cessation counseling)
  Interventions: Other: genotype-guided therapy; Behavioral: Smoking cessation counseling
- Standard (non-genotype guided) - NRT (Active Comparator): 1/2 of patients in this arm will be given nicotine replacement therapy (NRT; nicotine patch used according to FDA labeling) but this will NOT be based on the patient's genotype. Note that both nicotine replacement therapy and counseling are accepted treatments for smoking cessation in patients with coronary artery disease.
  Interventions: Drug: Nicotine patch
- Standard (non-genotype guided)- counseling (Active Comparator): 1/2 of patients in this arm will be given smoking cessation counseling but this will NOT be based on the patient's genotype. Note that both nicotine replacement therapy and counseling are accepted treatments for smoking cessation in patients with coronary artery disease.
  Interventions: Behavioral: Smoking cessation counseling

INTERVENTIONS:
Other: genotype-guided therapy — treatment based on patient's CHRNA5 rs16969968 genotype
  Arms: Genotype-guided (A allele carriers); Genotype-guided (GG homozygotes)
Drug: Nicotine patch
  Arms: Genotype-guided (A allele carriers); Standard (non-genotype guided) - NRT
Behavioral: Smoking cessation counseling
  Arms: Genotype-guided (GG homozygotes); Standard (non-genotype guided)- counseling

SUMMARY:
It has previously been shown that patients with coronary artery disease may have a harder time quitting smoking if they have a specific genetic profile and that these individuals have a better chance at quitting if they receive nicotine replacement therapy. The investigators hypothesize that determining which individuals with coronary artery disease should receive nicotine replacement therapy based on their genotype may improve the number of individuals who are able to quit smoking.This study randomizes treatment to that determined by the patient's genotype compared to standard, non-genotype-guided, treatment.

DETAILED DESCRIPTION:
In this study, the investigators propose to show the feasibility of incorporating genotype-guided therapy into post-MI smoking cessation therapy and/or smoking cessation therapy in patients with coronary artery disease (CAD) using the CHRNA5 rs16969968 variant as the pilot case. The investigators propose to genotype ½ of PRISM-GENOMICs patients who are active smokers within 48 hours of admission and to guide their smoking cessation therapy based on CHRNA5 rs16969968 genotype (A allele carriers will be given pharmacologic therapy and GG homozygotes will be given counseling). The investigators will use the other ½ as controls. The participants will be followed and the investigators will test whether the genotype-guided group has better rates of smoking cessation compared to the control group. This pilot study will lay the foundation for personalized, genotype-guided, post-MI therapy and/or therapy in patients with CAD.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* presenting to Barnes hospital cardiac catheterization laboratory with coronary artery disease or admitted to Barnes hospital within 24 hours of a type 1 myocardial infarction (heart attack)
* active smoker at time of presentation to Barnes Hospital
* participating in PRISM-GENOMICS observational study

Exclusion Criteria:

* Unable to provide informed consent
* Unable to answer questions (e.g. intubated)
* Incarcerated
* Complications of myocardial infarction (such as shock, hemodynamic instability, life- threatening infection, etc)
* Women of child-bearing age with positive pregnancy test or who is breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-07-21 (Actual); Primary Completion 2025-07-21 (Estimated); Study Completion 2025-07-21 (Estimated)

PRIMARY OUTCOMES:
Smoking Cessation | 1 month after enrollment
  Number of participants no longer smoking as assessed by telephone-administered questionnaire

SECONDARY OUTCOMES:
Smoking Cessation | 6 months after enrollment
  Number of participants no longer smoking as assessed by telephone-administered questionnaire
Smoking Cessation | 12 months after enrollment
  Number of participants no longer smoking as assessed by telephone-administered questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No